CLINICAL TRIAL: NCT00054249
Title: A Phase II Study Of Intravenous T900607-Sodium In Subjects With Previously Treated Gastric Carcinoma
Brief Title: T900607 in Treating Patients With Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Seidman Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TULA-T-607-006; CWRU-060214M; CDR0000269917 (Registry Identifier: PDQ (Physician Data Query)); TULA-TULI-1202
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2010-09

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — T 900607

INTERVENTIONS:
Drug: T900607

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of T900607 in treating patients who have gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (complete and partial) in patients with previously treated gastric or gastroesophageal junction carcinoma treated with T900607. (Gastric carcinoma closed to accrual as of 02/04.)
* Determine the duration of response and time to disease progression in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the safety profile of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive T900607 IV over 1 hour once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed gastric or gastroesophageal junction carcinoma (gastric carcinoma closed to accrual as of 02/04)
* Must have received 1 or 2 prior chemotherapy regimens for gastric carcinoma (gastric carcinoma closed to accrual as of 02/04)
* Bidimensionally measurable disease

  * At least 1 lesion that is at least 10 mm by CT scan
* No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3*
* Platelet count ≥ 100,000/mm^3*
* Hemoglobin ≥ 8.5 g/dL* NOTE: *Independent of growth factor or transfusion support

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* INR ≤ 1.5 (unless receiving anticoagulants)
* Albumin > 2.5 g/dL

Renal

* Creatinine ≤ 2 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease
* LVEF ≥ 50%
* No acute anginal symptoms

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* Able to comply with study procedures and follow-up
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No severe infection
* No other concurrent severe medical condition or comorbidity that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 7 days since prior growth factors or blood transfusions
* No concurrent therapeutic biological response modifier therapy
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy (including palliative radiotherapy)

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 4 weeks since prior investigational agents
* No other concurrent investigational anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2004-10 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Brell, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States